CLINICAL TRIAL: NCT06878794
Title: IIT Study on the Use of Medical Bio Glue for Repairing Meniscus Tears
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Ningbo University (Network)
Collaborators: The First Affiliated Hospital of Xinxiang Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-R049-03
Record Dates: First submitted 2024-11-28; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Unilateral Meniscus Tear of the Knee Joint
Keywords: Meniscus tear

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Sham Comparator): Using the meniscus suture system
  Interventions: Procedure: Using the meniscus suture system
- Experimental group (Active Comparator): Using medical biological glue for filling And Using the meniscus suture system
  Interventions: Combination Product: Using medical biological glue for filling And Using the meniscus suture system

INTERVENTIONS:
Combination Product: Using medical biological glue for filling And Using the meniscus suture system — Using medical biological glue for filling And Using the meniscus suture system
  Arms: Experimental group
Procedure: Using the meniscus suture system — Using the meniscus suture system
  Arms: Control group

SUMMARY:
To evaluate the safety and effectiveness of water triggered medical bioadhesive for meniscus tear repair

ELIGIBILITY:
Inclusion Criteria:

* 1. The patient is aged between 18 and 60 years old (including 18 and 60 years old), regardless of gender; 2. Unilateral meniscus tear of the knee joint; 3. Normal joint range of motion; 4. The subjects agree to participate in this trial and sign the "Subject Informed Consent Form".

Exclusion Criteria:

* 1. Body mass index BMI>32 kg/m2 (BMI=weight divided by height squared); 2. Patients with abnormal lower limb force lines that require correction; 3. Patients with multiple ligament injuries or complete meniscectomy; 4. Individuals with a history of allergies to biological glue as the chief complaint; 5. Patients with more than 2 or extensive cartilage defects in a single knee joint, and patients with bilateral knee joint cartilage defects; 6. Those who have undergone open knee surgery within the past 6 months; 7. Pregnant or lactating women, or those who plan to conceive during the trial period, and those whose blood HCG test results are positive before the trial; 8. Patients with infectious, immune, or metabolic arthritis in the knee joint; 9. Patients who participated in any other clinical trial or did not reach the trial endpoint within the first 3 months prior to enrollment; 10. Other circumstances determined by the researcher to be unsuitable for inclusion in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-25 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
MOCART score | Baseline (Before treatment), 6 and 12 months after treatment
Lysholm score | Baseline (Before treatment), 3、 6 and 12 months after treatment
IKDC score | Baseline (Before treatment), 3、 6 and 12 months after treatment

SECONDARY OUTCOMES:
T2 mapping | Baseline (Before treatment),12 months after treatment
Equipment use and evaluation | During operation
The occurrence of adverse events related to the test device | 12 months after treatment
The incidence of device related SAE requiring further surgical intervention within 12 months after surgical | 12 months after treatment
Equipment defect incidence rate | During operation

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Zhu, Study Chair — First Affiliated Hospital of Ningbo University
Locations (1):
- The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No